CLINICAL TRIAL: NCT04613947
Title: Investigation of the Effects of Consent Methods Performed According to Intelligence Types on Anxiety Associated with Third Molar Surgery
Brief Title: Effects of Consent Methods Performed According to Intelligence Types on Anxiety Associated with Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Dr. Damla Torul, Assistant Professor, Ordu University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2020/192
Record Dates: First submitted 2020-10-23; First posted 2020-11-03 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2022-12

CONDITIONS: Dental Anxiety
MeSH Terms: interventions — Informed Consent

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (Active Comparator): The group with standard (written and verbal) information without multiple intelligence test
  Interventions: Behavioral: Informed consent; Procedure: Third molar surgery
- Visual/Spatial: (Experimental): The group with higher visual intelligence according to the multiple intelligence test results and watch video. Also, will given with a written informed consent document
  Interventions: Behavioral: Informed consent; Procedure: Third molar surgery
- Verbal/Linguistic (Experimental): The group with higher verbal/linguistic intelligence according to the multiple intelligence test results and verbally informed in detail about the operation. lso, will given with a written informed consent document
  Interventions: Behavioral: Informed consent; Procedure: Third molar surgery
- Bodily/Kinesthetic (Experimental): The group with higher bodily/kinesthetic intelligence according to the multiple intelligence test results and informed with a dental model. lso, will given with a written informed consent document
  Interventions: Behavioral: Informed consent; Procedure: Third molar surgery

INTERVENTIONS:
Behavioral: Informed consent — The style of informing patients about the procedure they will undergo
Procedure: Third molar surgery — Surgical extraction of the third molar tooth

SUMMARY:
The aim of this study is to investigate the effect of information provided in accordance with intelligence type on anxiety associated with wisdom tooth surgery.

DETAILED DESCRIPTION:
The participants who will undergo third molar surgery divided into study and control groups. Study group divided further into three groups according to multiple intellegence test. Ultimately four groups created as follows;

1. Control: The group with standard (written and verbal) information without multiple intelligence test
2. Visual/Spatial: The group with higher visual intelligence according to the multiple intelligence test results and watch video. Also, will given with a written informed consent document.
3. Verbal/Linguistic: The group with higher verbal/linguistic intelligence according to the multiple intelligence test results and verbally informed in detail about the operation. lso, will given with a written informed consent document
4. Bodily/Kinesthetic: The group with higher bodily/kinesthetic intelligence according to the multiple intelligence test results and informed with a dental model. lso, will given with a written informed consent document To evaluate anxiety; participants will asked to complete MDAS questionnairre before and after consent, and after operation. Also, saliva samples will obtained to evaluate the salivary cortisol before and after consent, and after operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mandibular third molar tooth in vertical or mesioangular position according to Winter classification, class I and II ramus relationship according to Pell-Gregory classification and class B and C depth
* Patients who maintain their normal sleep patterns,
* Patients with ASA I status according to the American Society of Anesthesiologists (ASA) classification.

Exclusion Criteria:

* Patients did not agree to be a volunteer, and/or refused to watch videos or receive information in a different way from the standard procedure,
* Habits of Smoking and alcohol
* Patients who are pregnant or in the lactation period,
* Patients unable to cooperate,
* Patients having a psychiatric illness,
* Patients with systemic disease (local or systemic factors affecting salivary gland function, can cause changes in endocrine response)
* Patients using chronic medication and drugs that affect salivary cortisol levels, such as androgens, estrogens and corticosteroids.
* Patients with pericoronitis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Dental anxiety | at operation day (before and after operation and immediately after consent)
  Anxiety change being assessed with Modified Dental Anxiety Scale (MDAS) MDAS consists of five questions in total which measures anxiety at different stages of dental treatment. 1 (no anxious) to 5 (very anxious) options are available for each question. The sum of the scores varies from 5 to 25 and the values between 19-25 indicates high dental anxiety.

SECONDARY OUTCOMES:
Salivary cortisol level | at operation day (before and after operation and immediately after consent)
  The amount of cortisol in saliva samples

CONTACTS AND LOCATIONS:
Overall Officials: mehmet M ömezli, DDS PhD, Study Director — Ordu University; damla torul, DDS PhD, Principal Investigator — Ordu University
Locations (1):
- Ordu University, Ordu, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No